CLINICAL TRIAL: NCT06148688
Title: Effect of Digital Storytelling Intervention on Diabetes Self-Management in Pregnant Women With Gestational Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Izmir Katip Celebi University (Other)
Collaborators: Ege University (Other)
Responsible Party: Principal Investigator, Gulsen Isık, Research Assistant, Izmir Katip Celebi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21-2.1T/39
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy; Diabetes Self Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): In addition to the standard training, digital story videos were watched in the intervention group. Digital story videos created in line with four main topics related to diabetes self-management were sent to women via online platforms. During the follow-up period, reminder videos were sent once a week regarding the topics. Pre-test and post-test were administered face to face.
  Interventions: Other: Digital Story
- Control Group (No Intervention): The control group received only standard training.

INTERVENTIONS:
Other: Digital Story — Digital storytelling; It is used in education and training, business marketing, non-profit organizations such as libraries, community centers and museums, and health sciences education. Digital storytelling in health sciences can be a tool for patients and health science professionals to share their experiences, cope with diseases, and add a human element to health problems.
  In the study, digital stories were created to increase the self-management of pregnant women with gestational diabetes. In creating a digital story; Qualitative studies involving the self-management experiences of women with gestational diabetes have been examined in the literature. Using the results of the studies, scenarios were created that included factors that facilitate and complicate diabetes self-management. The created scenarios were used in the digital storytelling initiative. A total of four long and four short digital story videos were prepared.
  Arms: Intervention Group

SUMMARY:
The aim of this study is to evaluate the effect of digital storytelling intervention on diabetes self-management in women with gestational diabetes. It is a quasi-experimental study with a pretest-posttest control group.

The main hypotheses of the study are:

Digital storytelling has an impact on women with gestational diabetes' perception of diabetes self-management.

Digital storytelling has an impact on the diabetes self-efficacy levels of women with gestational diabetes.

DETAILED DESCRIPTION:
Women with gestational diabetes who apply to the obstetrics outpatient clinic of the hospital where the study is conducted or who have been hospitalized in the obstetrics clinic and who meet the inclusion criteria will be included in the study. As a result of the G-power analysis, the sample consisted of 21 interventions and 21 control groups. Pre-test data will be collected from pregnant women in both the control and intervention groups through scales.

In the hospital where the study was conducted, pregnant women with gestational diabetes are directed to the Endocrine outpatient clinic and receive standard training by the diabetes team. Pregnant women in the intervention group will be shown videos created in addition to the standard training of the institution where the research data were collected.

Pregnant women in the intervention group will be shown videos created in addition to the standard training of the institution where the research data were collected. Pregnant women participating in the study will be followed for four weeks. Pre-test data will be collected from pregnant women who meet the sampling criteria within the first week and how the research will proceed will be explained. Four separate videos, created specifically for each determined topic, will be sent to women daily via online environments during the first week and they will be made available for viewing. Once a week, short videos will be sent to the pregnant woman as a reminder and she will be allowed to watch them. Women will be asked to keep records of their blood sugar monitoring results for four weeks. In the fourth week, post-test data from women will be collected through scales.

Scales to be used in the research

* Introductory Information Form (pre-test)
* Diabetes Self-Efficacy Scale (pre-test/post-test)
* Perceived Diabetes Self-Management Scale (pre-test/post-test)
* International Physical Activity Questionnaire (pre-test/post-test)
* Blood Sugar Monitoring Form (post-test)

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older
* Being diagnosed with Gestational Diabetes
* 24-32. being between weeks of pregnancy
* Having a treatment plan made after gestational diabetes diagnosis
* Volunteering to participate in the study
* Knowing how to read and write Turkish
* Not having any pregnancy complications other than Gestational Diabetes
* Having a smart phone

Exclusion Criteria:

-Pregnant women who do not meet the inclusion criteria will be excluded from the study. Moreover; Pregnant women whose blood sugar monitoring was terminated by the doctor during the follow-up, who did not continue hospital checks during the research period or could not be reached, and who experienced preterm labor before the end of the follow-up will be excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Perceived Diabetes Self-Management Scale | before and end of the interventions (fourth weeks)
  The Turkish adaptation of the scale, which was adapted and validated by Wallston et al. (2007), was made by Bayındır Çevik (2010).The scale consists of 7 items and is of 5-point likert type.A high total score indicates that the individual's awareness of diabetes management is very good.
Diabetes Self-Efficacy Scale | before and end of the interventions (fourth weeks)
  This scale was developed by Lorig et al. in 2009 to determine the self-efficacy of individuals with diabetes and was adapted into Turkish by Mankan et al. in 2017.The Likert type scale consists of 8 items. The items of the scale have a numbering system between 1 and 10 (1-I do not feel safe at all, 10-I am completely confident).The scale has no cut-off point. As individuals' total scale scores increase, their self-efficacy also increases.
International Physical Activity Questionnaire | before and end of the interventions (fourth weeks)
  The International Physical Activity Questionnaire was designed to detect the physical activity and sedentary lifestyles of adults. Craig et al. (2003) and the Turkish validity and reliability of the questionnaire developed by Öztürk (2005). The questionnaire is recommended for adults aged 18-69. The short-form questionnaire consists of four separate sections and a total of seven questions. The questionnaire includes questions about physical activity performed for at least 10 minutes in the last seven days.
  Calculation of the total score of the short form includes the sum of the duration (minutes) and frequency (days) of walking, moderate activity and vigorous activity. From these calculations, a score in MET-minutes is obtained. One MET-minute; It is calculated by multiplying the minutes of activity performed by the MET score. Walk = 3.3 METs, Moderate physical activity = 4.0 METs, Vigorous physical activity = 8.0 METs

SECONDARY OUTCOMES:
Blood Sugar Monitoring Form | first week, second week, third week and fourth week
  Women in the sample group will be asked to record their fasting and 1-hour postprandial blood sugar results in the morning, noon and evening for 4 weeks. The blood sugar monitoring form was prepared by the researcher.

CONTACTS AND LOCATIONS:
Overall Officials: Gülşen Işık, Principal Investigator — Izmir Katip Celebi University
Locations (1):
- Izmir Katip Celebi University, Çiğli, İzmir, Turkey (Türkiye)